CLINICAL TRIAL: NCT05038280
Title: Let´s Talk About Children Intervention in a School Context
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Lotta Allemand, Principal Investigator, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: University of Helsinki
Record Dates: First submitted 2021-08-24; First posted 2021-09-09 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Children's Wellbeing; Child Overall Health Related Quality of Life; Burnout
Keywords: Let's Talk about Children; School; Teacher-Student Relationship; Teacher-Parent Relationship; Children's Wellbeing; Teachers' Occupational Wellbeing; Parental Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Let's Talk about Children intervention (Experimental): Teachers, students, and parents in Finland, that take part in the LTC -intervention.
  Interventions: Behavioral: Let's Talk about Children intervention
- Control group (No Intervention): The control group includes teachers who do not use the method in their work and students and parents who do not participate in the discussions.

INTERVENTIONS:
Behavioral: Let's Talk about Children intervention — The LTC -intervention includes two steps: Let´s Talk about Children discussion and Let´s Talk about Children network meeting. Students, students´ parents, and a teacher take part in the LTC -discussion. The LTC logbook is used as the framework for the discussions. The LTC discussion depicts the child's ordinary day in all developmental contexts and an action plan is made with parents to enhance the identified strengths and to give support in vulnerabilities. When the action plan is difficult to carry out without further participants, the LTC-Network meeting is planned with parents (and sometimes also the child). LTC-Network meeting provides a forum for case-based cross-sectoral collaboration, including also the families and their social network.
  Arms: Let's Talk about Children intervention

SUMMARY:
The aim of this study is to examine the fidelity, the perceived benefits, and the effectiveness of the Let's Talk about Children (LTC) -intervention in a school context. The Let's Talk about Children method is a standardised, family-focused intervention aimed to build a shared understanding between parents, children, and teachers to find ways of working together to support the child's everyday life, well-being, learning, and development, both at home and at school. The Let's Talk about Children intervention is used in several different schools in Finland. The study examines the effects of the Let's Talk about Children method on the teacher-student relationship, the trust between teachers and parents and the students', teachers' and parents' well-being. Participants (N=1316 school-children, N=188 school-teachers and N=1316 parents) are recruited and divided into intervention and control groups. The intervention group consists of teachers who use the Let's Talk about Children method in their work and those students and parents who participate in the Let's Talk about Children discussions. The control group includes teachers who do not use the method in their work and students and parents who do not participate in the discussions. The fidelity and perceived benefits of the method are examined in the intervention group. Otherwise, there is two data collection points. The data is collected in intervention and control groups before the intervention and 6 months after the intervention.

DETAILED DESCRIPTION:
The Let´s Talk about Children Intervention method is one of the Effective Child & Family Methods. The LTC -method was developed as a part of the Functioning Child & Family project co-ordinated by the Finnish Institute for Health and Welfare. The LTC -intervention includes two steps: Let´s Talk about Children discussion and Let´s Talk about Children network meeting. The method is used in social- and healthcare services, kindergartens and schools but has been studied mainly in the field of social- and healthcare services. The aim of the LTC -work in schools is to support the child's well-being, learning and development in everyday life. The other aim of the LTC -intervention in the school environment is to support teachers and parents in their everyday interactions and activities with children. The LTC is used to build a common comprehensive understanding of the child and his/her situation in school and at home, and to plan actions based on this understanding. The aim is also to build a mutually supportive parent-teacher relationship based on respect. Students, parents and a teacher take part in the discussion. The LTC logbook is used as the framework for the discussions. The LTC -method is based on an ecological, transactional model of child development.

The research questions of the research study are:

Is the intervention delivered as designed? How do teachers/parents experience the Let´s Talk about Children intervention? Does the Let´s Talk about Children intervention have an effect on teacher and student relationship? Does the Let´s Talk about Children intervention have an effect on teacher and parent relationship? Does the Let´s Talk about Children intervention have an effect on students´ well-being? Does the Let´s Talk about Children intervention have an effect on teachers´ well-being at work? Does the Let´s Talk about Children intervention have an effect on parents´ well-being?

ELIGIBILITY:
Inclusion Criteria:

* First-grade students
* Students' parents
* First-grade teachers
* Sufficient Finnish language skills

Exclusion Criteria:

- Insufficient Finnish language skills

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in teacher and parent relationship | 6 months after baseline
  A set of teacher-parent interaction tests
Change in children's wellbeing: psychiatric symptoms | 6 months after baseline
  SDQ - The Strengths and Difficulties Questionnaires. The SDQ has 25 items and consists of sub-scales to measure emotional symptoms, conduct problems, hyperactivity/inattention, peer problems and prosocial behavior. Scoring 0-40 (prosocial scale is not included in the total score), higher score meaning more problems.
Change in children's wellbeing: health-related quality of life | 6 months after baseline
  The Kid-KINDL-R. The KINDL questionnaire is a generic instrument for assessing Health-Related Quality of Life in children and adolescents aged 3-17. The KINDLR questionnaire consists of 24 Likert-scaled items associated with six dimensions: physical well-being, emotional well-being, self-esteem, family, friends and everyday functioning (school or nursery school/kindergarten). The sub-scales of these six dimensions can be combined to produce a total score. The total score is transformed to a scale of 0-100 such that higher score represents a better outcome, i.e. better HRQoL.
Change in teacher and student relationship | 6 months after baseline
  Student-Teacher Relationship Scale (short form). The STRS is a teacher-report instrument designed for teachers of children between the ages of 3 and 12 which measures a teacher's perception of conflict, closeness, and dependency with a specific child. Teachers will complete the Student-Teacher Relationship Scale (short form) for each child in his/her classroom to assess Student-Teacher closeness and Student-Teacher conflict. Seven items make up the Closeness subscale, 8 items make up the Conflict subscale. Teachers respond to each item on a five-point scale (1 = definitely does not apply to 5 = definitely applies), with higher scores indicating a better outcome for the closeness scale and a worse outcome for the conflict scale.

SECONDARY OUTCOMES:
Change in teachers' occupational wellbeing: burnout | 6 months after baseline
  Bergen Burnout Indicator 15. The Bergen Burnout Inventory is comprised of 15 items, ranging from 1 to 5. The total score range is from 15 to 75 with a higher score reflecting higher burnout.
Change in teachers' occupational wellbeing: job engagement | 6 months after baseline
  The Utrecht Work Engagement scale. The UWES is comprised of 9 items, ranging from 1 to 5. The total score range is from 9 to 45 with a higher score indicating more work engagement.
Change in parents' wellbeing: burnout | 6 months after baseline
  Parental Burnout Assessment (Finnish version of the PBA). The scale consists of 23 items. Nine measure exhaustion in one's parental role, six measure contrast with the previous parental self, five measure feelings of being fed up as a parent and three measure emotional distancing from one's children. All item are rated on a 7-point Likert scale (0 = never; 6 = daily).

CONTACTS AND LOCATIONS:
Overall Officials: Lotta Allemand, Principal Investigator — University of Helsinki
Locations (1):
- University of Helsinki: Faculty of Educational Sciences, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allemand L, Niemela M, Merikukka M, Salmela-Aro K. The "Let's Talk about Children" intervention in a Finnish school context: fidelity, parents' experiences, and perceived benefits. Front Psychol. 2023 Jun 9;14:1183704. doi: 10.3389/fpsyg.2023.1183704. eCollection 2023. PMID 37359866